CLINICAL TRIAL: NCT04939506
Title: COVID-19 Vaccine Education at the Point of Testing to Increase Vaccine Uptake in Vulnerable Communities in Southeastern Louisiana
Brief Title: COVID-19 Vaccine Education at the Point of Testing to Increase Vaccine Uptake in Vulnerable Communities in SE Louisiana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xavier University of Louisiana. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB850-21
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Covid19; Vaccine Refusal; Vaccine Hesitancy
Keywords: Vaccine Completion; COVID19 Testing; COVID19 Education; Point of Care Testing; Healthcare Personnel Education; Healthcare Disparities
MeSH Terms: conditions — COVID-19; Vaccination Refusal; Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants Which Receive COVID-19 Vaccine Education at the Point of COVID-19 Testing (Experimental): Vaccine education will be focused on addressing misinformation and concerns in a culturally competent manner with referral to resources. The vaccine education model will be translated to reach minority groups including African Americans, Vietnamese Americans and Hispanic Americans.
  Interventions: Behavioral: COVID-19 Vaccine Education at the Point of COVID-19 Testing

INTERVENTIONS:
Behavioral: COVID-19 Vaccine Education at the Point of COVID-19 Testing — A rapid vaccination education model to be delivered at the point of COVID-19 testing by pharmacy students, pharmacy technicians, nurse's aides and other health care personnel. The intervention will include: 1) 15 minute vaccine counseling, 2) print material 3) referral to a dedicated vaccine website with feedback forums and 4) opportunity to sign-up for one-on-one vaccine counseling with a clinical pharmacist

SUMMARY:
This project is a 2-year study to investigate vaccine hesitancy and vaccine completion among vulnerable communities in the Southeastern Louisiana region. This study will be used to track COVID-19 vaccine completion among patients who seek testing, either as in-person or purchasing at home COVID testing, from pharmacies, urgent cares and clinics using a rapid vaccine education model delivered at the point of care.

DETAILED DESCRIPTION:
This project is a 2-year study to investigate vaccine hesitancy and vaccine completion among vulnerable communities in the Southeastern Louisiana region. This study will be used to track COVID-19 vaccine completion among patients who seek testing, either as in-person or purchasing at home COVID testing, from pharmacies, urgent cares and clinics. The proposal will introduce a rapid vaccination education model to be delivered at the point of COVID-19 testing by pharmacy students, pharmacy technicians, nurse's aides and other health care personnel and includes monitoring for COVID-19 vaccine completion among enrolled patients. Investigators anticipate an increase in COVID-19 vaccine completion rates for those who participate in the rapid vaccination education model.

ELIGIBILITY:
Inclusion Criteria:

* Unvaccinated adult participants, 18-99 years of age, able to provide informed consent, and to communicate in English, Spanish or Arabic. Also, individuals with incomplete vaccination (primary series or COVID-19 booster).

Exclusion Criteria:

* Persons fully vaccinated for COVID-19 (including primary series and boosters), persons with any documented allergies to components of the COVID-19 vaccines, or contraindications to receiving a COVID-19 vaccine.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
COVID-19 Vaccine Completion | 9 months intervention
  COVID-19 vaccination verified by the Louisiana Links© system

SECONDARY OUTCOMES:
Vaccine Hesitancy Likelihood Scale | 9 months post intervention
  Measured on a 5-point scale indicating likelihood to be vaccinated. The scale ranges from 1 (Not at all likely to be vaccinated), 2 (Not likely to be vaccinated), 3 (No opinion/Undecided about vaccination), 4 (Likely to be vaccinated) to 5 (Very likely to be vaccinated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Al-Dahir, PharmD, Principal Investigator — Xavier University of Louisiana.; Klaus Heyer, PhD, Principal Investigator — Nunez Community College
Locations (1):
- Xavier University of Louisiana, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No